CLINICAL TRIAL: NCT07148180
Title: A Multi-Site Break Through Cancer Trial: Targeting Measurable Residual Disease in Patients With Acute Myeloid Leukemia: A Phase 1/2 Study of Tagraxofusp, Azacitidine, and Venetoclax
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jacqueline Garcia, MD (Other)
Collaborators: Stemline Therapeutics, Inc. (Industry); Break Through Cancer Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Jacqueline Garcia, MD, Sponsor-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25-330
Record Dates: First submitted 2025-08-20; First posted 2025-08-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukaemia (AML); Leukemia; Blood Cancer; Blood Cancers
Keywords: Acute Myeloid Leukemia; AML; Measurable Residual Disease; Myeloid Neoplasms; Blood Cancer; Blood Cancers
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Hematologic Neoplasms; Neoplasm, Residual | interventions — tagraxofusp; Azacitidine; venetoclax

STUDY DESIGN:
Intervention Model Description: The study includes a phase 1 dose-escalation phase to determine the MTD and RP2D, followed by a phase 2 dose-expansion phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Phase 1 Dose Escalation (Experimental): Up to 12 participants will be enrolled in a standard 3+3 design to determine the maximum tolerated dose/RP2D for Tagraxofusp in combination with azacitidine and venetoclax starting at Dose Level 1 and escalating to Dose Level 2 according to dose-limiting toxicity rules.
  * Baseline visit
  * Cycles 1 through 2 (28 day cycles):
    * Days 1 through 7: Predetermined dose of Azacitidine 1x daily.
    * Days 4 through 6: Predetermined dose of Tagraxofusp 1x daily.
    * Days 1 and 14: Predetermined dose of Venetoclax 1x daily
    * Day 28: bone marrow aspiration and biopsy
  * Cycles 3 through 24 (28 day cycles):
    * Days 1 through 7: Predetermined dose of Azacitidine 1x daily.
    * Days 4 through 6: Predetermined dose of Tagraxofusp 1x daily.
    * Days 1 and 14: Predetermined dose of Venetoclax 1x daily
  * Bone marrow aspirations/biopsies on Day 1 of Cycles 4, 6, 9, 12, and then every 3 cycles.
  * End of treatment visit with bone marrow aspiration and biopsy
  * Follow up for up to 2 years
  Interventions: Drug: Tagraxofusp; Drug: Azacitidine (AZA); Drug: Venetoclax
- Arm 2: Phase 2 Dose Expansion (Experimental): 19 Participants will receive Tagraxofusp at the RP2D in combination with Azacitidine and Venetoclax and will complete:
  * Baseline visit
  * Cycles 1 through 2 (28 day cycles):
    * Days 1 through 7: Predetermined dose of Azacitidine 1x daily.
    * Days 4 through 6: Predetermined dose of Tagraxofusp 1x daily.
    * Days 1 and 14: Predetermined dose of Venetoclax 1x daily
    * Day 28: bone marrow aspiration and biopsy
  * Cycles 3 through 24 (28 day cycles):
    * Days 1 through 7: Predetermined dose of Azacitidine 1x daily.
    * Days 4 through 6: Predetermined dose of Tagraxofusp 1x daily.
    * Days 1 and 14: Predetermined dose of Venetoclax 1x daily
  * Bone marrow aspirations/biopsies on Day 1 of Cycles 4, 6, 9, 12, and then every 3 cycles.
  * End of treatment visit with bone marrow aspiration and biopsy
  * Follow up for up to 2 years
  Interventions: Drug: Tagraxofusp; Drug: Azacitidine (AZA); Drug: Venetoclax

INTERVENTIONS:
Drug: Tagraxofusp — A CD123-directed cytotoxin, Single-use vial, via intravenous (into the vein) infusion per protocol.
  Other Names: ELZONRIS; SL-401
Drug: Azacitidine (AZA) — A cytidine nucleoside analog, single-use vial, via intravenous infusion or subcutaneous (under the skin) injection per standard of care.
  Other Names: VIDAZA; Onureg
Drug: Venetoclax — A BCL-2 inhibitor, tablet, via orally per standard of care.
  Other Names: VENCLEXTA; C45H50ClN7O7S

SUMMARY:
The purpose of this research study is to test the safety and efficacy of a new drug combination with three agents, azacitidine, venetoclax and tagraxofusp. Leftover (residual) leukemia disease that is not visible by eye can be increase the chance of disease recurrence. This research study is to determine if the combination therapy can safely help to control residual Acute Myeloid Leukemia (AML) and to prevent disease recurrence.

The names of the study drugs involved in this study are:

* Tagraxofusp (a type of CD123-directed cytotoxin)
* Azacitidine (a type of standard of care cytidine nucleoside analog)
* Venetoclax (a type of standard of care BCL-2 inhibitor)

DETAILED DESCRIPTION:
This phase 1/2 study, single-arm, multi-center, open-labeled clinical trial is to test the safety and efficacy of a new drug combination with three agents, azacitidine, venetoclax and tagraxofusp. Leftover (residual) leukemia disease that is not visible by eye can be increase the chance of disease recurrence. This research study is to determine if the combination therapy can safely help to control residual Acute Myeloid Leukemia (AML) and to prevent disease recurrence.

A Phase 1/2 clinical trial tests the safety and effectiveness of an investigational drug combination to learn whether the drug combination works in treating a specific disease. The Phase 1 safety run-in part of the study will determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) for tagraxofusp in combination with Azacitidine and Venetoclax. Phase 2 will test the RP2D for Tagraxofusp in combination with azacitidine and venetoclax.

The U.S. Food and Drug Administration (FDA) has approved the doublet combination of venetoclax and azacitidine for the treatment of AML.

The U. S. FDA has approved Tagraxofusp monotherapy as a therapy for another type of leukemia called blastic plasmacytoid dendritic cell neoplasm.

The U.S. Food and Drug Administration (FDA) has not approved the combination of azacitidine, venetoclax and tagraxofusp as a treatment for AML.

The research study procedures include screening for eligibility, in-clinic visits, blood tests, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, or Positron Emission (PET) scans, X-rays, echocardiograms (ECGs), electrocardiograms (EKGs), and bone marrow biopsies and aspirations.

Participation in this research study is expected to last about 4 years.

It is expected that about 31 people will take part in this research study.

Stemline Therapeutics is supplying the study drug, Tagraxofusp. Break Through Cancer is providing funding to support the laboratory services.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* History of known diagnosis of Acute Myeloid Leukemia (including de novo, secondary or AML arising from MDS).
* Subjects must be in CR, CRi, or CRh with <5% morphologic blasts in bone marrow
* Any evidence of CD123+ by central assessment.
* Participants must have measurable disease, defined as ≥ 0.1% by multiparametric flow cytometric assay as assessed by central laboratory
* ECOG performance status ≤2 (see Appendix A).
* Subjects must have adequate organ and marrow function as defined below:

  * total bilirubin ≤ 1.5 x institutional upper limit of normal unless due to Gilbert or non-hepatic in origin
  * AST(SGOT) and ALT(SGPT) ≤ 3.0 × institutional upper limit of normal
  * Creatinine clearance ≥ 45 ml/min GFR by MDRD
* Albumin ≥ 3.2 g/dL
* Left ventricular ejection fraction ≥ institutional lower limit of normal by MUGA or echocardiogram within 30 days of first protocol treatment. This can be locally assessed.
* Pregnancy potential: Female subjects of childbearing potential must have negative results for pregnancy test. Females with reproductive potential are advised to use effective contraception during study treatment and for at least 6 months after last dose. Similarly, males with female partners of reproductive potential are advised to use effective contraception during treatment and for at least 3 months after the last dose. Men must agree to abstain from donating sperm.
* Subject is able and willing to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Prior treatment with CD123-targeted therapy
* Known diagnosis of acute promyelocytic leukemia.
* Subjects who received intensive anti-leukemic chemotherapy within 2 weeks from first dose of study. If on venetoclax, subjects must be off venetoclax for at least 5 days
* Subjects pre-arranged for SCT are only excluded if it is imminent.
* History of prior allogeneic stem cell transplant
* Subject has uncontrolled, clinically significant pulmonary disease (e.g. COPD, pulmonary hypertension, etc.) that in the opinion of the Investigator would put the subject at significant risk for pulmonary complications during the study.
* Subject has experienced Grade 3 or Grade 4 capillary leak syndrome (CLS) in the past for any reason
* Subjects with known HBV and/or HCV infection must have undetectable viral load during screening (HBV and HCV testing are not required.) Participants with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative-, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate.
* Subjects with known HIV positivity are permitted provided they have undetectable viral load at the time of screening (HIV testing is not required).
* Subject has a concurrent malignancy or prior malignancy within the 6-month period before screening. To be eligible, subjects must be in remission from the prior malignancy at least 6 months prior to screening and all treatment-related toxicities must have resolved to ≤ Grade 1 except for alopecia. Exceptions include adequately treated basal or squamous cell skin cancer, superficial bladder cancer, adequately treated carcinoma in situ of the cervix or uterus, or carcinoma in situ of the breast, previous malignancy confined and surgically resected (or successfully treated with other modalities) with curative intent, which are permissible for inclusion. Maintenance therapy, hormonal therapy, or steroid therapy for a well-controlled concurrent malignancy is allowed.
* Subject has uncontrolled systemic fungal, bacterial, or viral infection, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antivirals, or antifungals, either IV or oral. However, subjects with controlled infection still requiring anti-infectives are eligible.
* Subjects with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, that have New York Heart Association Functional Class III or IV symptoms.
* Subject has evidence of ongoing alcohol or drug abuse
* Subjects with known active/symptomatic CNS involvement. CNS prophylaxis allowed
* Subjects receiving moderate or strong P450 3A (CYP3A) inducers within 7 days of start of study therapy. See Appendix B for examples
* Subjects with uncontrolled intercurrent illness.
* Administration or consumption of any of the following within 3 days prior to the first dose of study drug:

  * grapefruit or grapefruit products
  * Seville oranges (including marmalade containing Seville oranges)
  * star fruit
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with trial therapy, breastfeeding should be discontinued if the mother is treated on trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) of tagraxofusp in combination with fixed dose of Azacitidine and Venetoclax [Phase I] | Up to 28 days
  Definition of RP2D is outlined in protocol section 5.4.
Number of Participants Experienced Dose-Limiting Toxicity (DLT) [Phase I] | Up to 28 days
  Definition of Dose Limiting Toxicity (DLT) is outlined in protocol section 5.4.
Measurable Residual Disease (MRD) conversion rate [Phase II] | Up to 4 months
  MRD conversion rate is defined as the proportion of participants that achieve multi-parametric flow cytometry (MFC) MRD conversion (positive to negative) within the first four cycles of therapy. MRD negativity will be defined according to 2021 ELN MRD Working Party Consensus Guidelines and central lab MRD will be used to make this determination: CR with negative MFC-MRD negative refers to achievement of flow MRD negativity: MFC-MRD negative in bone marrow defined as <0.1% (same as <10^-3).

SECONDARY OUTCOMES:
Duration of Remission (DOR) | Disease response assessments will be conducted at baseline, day 1 of cycles 2, 4, 6, 9, and 12, then every 3 cycles thereafter during treatment, and at end of treatment (2 years) or upon suspected relapse. Each cycle is 28 days.
  DOR based on Kaplan-Meier method is measured from the time criteria are met for complete remission (CR) and partial remission (PR) until the first data that recurrent or disease progression. Response criteria is listed in Appendix D.
Median Overall Survival (OS) | Participants off protocol treatment but remaining on study will have survival status assessed every 12 weeks for up to 2 years. Maximum treatment duration is 2 years.
  Overall Survival (OS) based on Kaplan-Meier method is defined as the time from study treatment to death due to any cause or censored at date last known alive. All surviving participants will be censored at time of final follow up.
Median Relapse-free survival (RFS) | Disease response assessments will be conducted at baseline, day 1 of cycles 2, 4, 6, 9, and 12, then every 3 cycles thereafter during treatment, and at end of treatment (2 years) or upon suspected relapse. Each cycle is 28 days.
  Relapse-Free Survival (RFS) is defined as the time from study treatment to evidence of relapse (morphologic relapse per ELN 2022 criteria) or at death due to any cause including underlying disease. Participants alive without disease progression are censored at date of last follow up.
Median Event-free Survival (EFS) | Disease response assessments will be conducted at baseline, day 1 of cycles 2, 4, 6, 9, and 12, then every 3 cycles thereafter during treatment, and at end of treatment (2 years) or upon suspected relapse. Each cycle is 28 days.
  Event-free survival is defined as the number of days from the date of treatment initiation (i.e., C1D1) to the date of documented treatment failure, relapse (MRD or morphologic), progression, or death from any cause, whichever occurs first, and will be calculated for all participants. If neither disease progression nor death is documented prior to study termination, analysis cutoff, or the start of confounding anticancer therapy, these endpoints will be censored at the date of last tumor assessment date.
Bridge to Transplantation Rate | Maximum treatment duration is 2 years.
  Bridge to transplantation rate is defined as the proportion of participants that are eligible for transplant that then undergo transplant after this study treatment
Cumulative Incidence of Relapse Participants (including morphologic relapse and MRD relapse) | Maximum treatment duration is 2 years.
  The number of participants who experienced either morphologic relapse (≥5% blasts in bone marrow by morphology or emergence of leukemic blasts in peripheral blood while on study treatment) or MRD relapse (flow MRD ≥0.1% after achievement of flow MRD <0.1% on trial treatment while on study treatment).
Capillary Leak Syndrome and Febrile Neutropenia Rate | Adverse events will be collected while participants receive study treatment. Maximum treatment duration is 2 years.
  "Capillary leak syndrome and febrile neutropenia rate is defined as the number of participants who experience capillary leak syndrome or febrile neutropenia on treatment. Toxicities will be graded according to the NCI CTCAE, V5.0 as reported on case report forms.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Garcia, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu